CLINICAL TRIAL: NCT04607252
Title: Comparing Metformin Plus Megestrol Acetate with Megestrol Acetate Alone As a Fertility-sparing Treatment in Patients with Atypical Endometrial Hyperplasia
Brief Title: Metformin Plus Megestrol Acetate As a Fertility-sparing Treatment in Patients with Atypical Endometrial Hyperplasia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Our clinical trial NCT03241888 showed LNG-IUS had a better treatment efficacy than Megestrol Acetate (MA) alone. The median CR time for MA group, LNG-IUS group and MA plus LNG-IUS group was 7.0±0.3 months, 4.4±1.0 months and 5.7±1.2 months.
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Prof.Dr, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V01 2020-10
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Atypical Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Metformin; Megestrol Acetate

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin plus megestrol acetate (Experimental): Metformin 1500mg per day plus megestrol acetate 160mg per day.
  Interventions: Drug: Metformin plus Megestrol acetate
- Megestrol acetate (Active Comparator): Megestrol acetate 160mg per day.
  Interventions: Drug: Megestrol Acetate

INTERVENTIONS:
Drug: Metformin plus Megestrol acetate — metformin 1500mg, per day, oral; megestrol acetate 160mg per day, oral
  Arms: Metformin plus megestrol acetate
Drug: Megestrol Acetate — megestrol acetate 160mg per day, oral
  Arms: Megestrol acetate

SUMMARY:
To verify whether metformin could improve the effect of progestin as fertility-sparing treatment in patients with atypical endometrial hyperplasia(AEH).

DETAILED DESCRIPTION:
Whether metformin could improve the effect of progestin as fertility-sparing treatment in patients with atypical endometrial hyperplasia(AEH) is still not clear. Our previous finding from subgroup analysis in a phase II randomized controlled trial showed that 39.6% of AEH patients in metformin plus megestrol acetate group achieved complete response, compared with 20.4% in group of megestrol acetate alone. This trial aim to fully testify the effect of metformin in fertility-sparing treatment for AEH patients with adequate sample size.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years old;
2. pathologically diagnosed with AEH for the first time;
3. desire to preserve their fertility;
4. no signs of suspicious myometrial invasion or extrauterine metastasis by enhanced magnetic resonance imaging (MRI), enhanced computed tomography (CT) or transvaginal ultrasonography (TVUS);
5. no contraindication for metformin, megestrol acetate or pregnancy;
6. no hormone or metformin treatment within 6 months before entering the trial;
7. not pregnant when participating in the trial;
8. willing to follow the trial arrangement after being fully informed of all the risks and inconveniences caused by the trial.

Exclusion Criteria:

Patients who had one or more of the following conditions:

1. allergy history or contraindications for megestrol acetate or metformin;
2. pregnant when initiating the study;
3. alcoholism, severe infection, severe chronical diseases (dysfunction of heart, liver, lung or kidney);
4. high risk of thrombosis;
5. recurrent AEH;
6. endometrial cancer;
7. other malignancy history.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Complete response within 16 weeks of treatment | 16 weeks
  reversion of AEH The reversion of AEH to proliferative or secretory endometrium

SECONDARY OUTCOMES:
Complete response within 32 weeks of treatment | 32 weeks
  The reversion of AEH to proliferative or secretory endometrium
Adverse events | 32 weeks
  Adverse events during the treatment of metformin plus megestrol acetate or megestrol acetate alone
2-year recurrence rate | 2 years
  recurrence rate within 2 years after the treatment
2-year pregnancy rate | 2 years
  Pregnancy rate within 2 years after the treatment
2-year live-birth rate | 2 years
  Live-birth rate within 2 years after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Chen, PHD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data will be shared with other researchers without patients' personal information after all the findings being published.